CLINICAL TRIAL: NCT04946513
Title: The Influence of Hip Arthroscopy on Postoperative Muscle Volumes in Patients With Femoroacetabular Impingement Syndrome
Brief Title: Hip Arthroscopy Improves Muscle Volumes in Patients With Femoroacetabular Impingement Syndrome
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019451
Record Dates: First submitted 2021-06-27; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Femoroacetabular Impingement Syndrome
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients with femoroacetabular impingement syndrome and underwent hip arthroscopy。
  Interventions: Other: Muscle volumes were measured on pre- and postoperative MRI scans.

INTERVENTIONS:
Other: Muscle volumes were measured on pre- and postoperative MRI scans. — Muscle volumes were measured on pre- and postoperative MRI scans.

SUMMARY:
To explore the changes of the muscles around the hip joint after hip arthroscopy for patients with femoral acetabular impingement syndrome.

DETAILED DESCRIPTION:
Retrospectively investigate the influence of hip arthroscopy on the muscle volume around the hip joint, and to provide important information for clinicians to make diagnosis and treatment plan of hip joint disease.

ELIGIBILITY:
Inclusion Criteria: (1) Age 18-50 years old; (2) Diagnosed femoroacetabular impingement syndrome; (3) Conservative treatment ineffective; (4) complete preoperative and postoperative MRI images; -

Exclusion Criteria: (1) bilateral; (2) revision; (3) osteoarthritis; (4) acetabular dysplasia; (5) history of hip and knee joint disease or surgery; (6) femoral head necrosis; (7) sacroiliac joint disease.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with femoroacetabular impingement syndrome and underwent hip arthroscopy.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Muscle volumes | 1 year after hip arthroscopy
  Difference between pre- and postoperative muscle volumes

CONTACTS AND LOCATIONS:
Overall Officials: Jian-quan Wang, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No